CLINICAL TRIAL: NCT02888925
Title: Evaluation of Neuropsychological Effects of Drug-resistant Anterior Temporal Epilepsy and Anterior Temporal Lobectomy in Face Perception
Brief Title: Anterior Temporal Epilepsy Neuropsychological Assessment of Faces
Acronym: ATENA-F
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013-A00515-40
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Anterior Temporal Epilepsy; Anterior Temporal Lobectomy; Face Perception
MeSH Terms: interventions — Anterior Temporal Lobectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epilepsy (Other): Patients do face specific tests during conventional pre-lobectomy intercritical assessment hospitalization (inclusion, day 0) and after 6 and 18 months from anterior temporal lobectomy
  Interventions: Other: Mooney test; Other: Benton Face Recognition test; Other: Face inversion effect test; Other: Face composite effect test; Other: Cambridge Face Memory Test; Other: Matching different view test; Other: Memorizing and recognition of new faces test; Other: Memorizing and recognition of new objects test; Other: Recognition of celebrities and access to semantic information test; Procedure: Lobectomy
- Control (Other): Control individuals do face specific tests during inclusion visit (day 0) and after X months (X = time from day 0 and lobectomy of matched patient + 6 months)
  Interventions: Other: Mooney test; Other: Benton Face Recognition test; Other: Face inversion effect test; Other: Face composite effect test; Other: Cambridge Face Memory Test; Other: Matching different view test; Other: Memorizing and recognition of new faces test; Other: Memorizing and recognition of new objects test; Other: Recognition of celebrities and access to semantic information test

INTERVENTIONS:
Other: Mooney test
Other: Benton Face Recognition test
Other: Face inversion effect test
Other: Face composite effect test
Other: Cambridge Face Memory Test
Other: Matching different view test
Other: Memorizing and recognition of new faces test
Other: Memorizing and recognition of new objects test
Other: Recognition of celebrities and access to semantic information test
Procedure: Lobectomy — In patients with anterior temporal epilepsy, at 6 to 12 months after inclusion, depending on surgery decision taken after pre-surgery conventional intercritical assessment
  Arms: Epilepsy

SUMMARY:
The purpose is to evaluate neuropsychological effects of anterior temporal epilepsy in face perception by comparison of performances of epileptic patients and control individuals, sex-, age- and socio-educational level-matched.

Secondary purposes are to prospectively evaluate neuropsychological impact of anterior temporal lobectomy performed for surgical treatment of anterior temporal epilepsy on face perception (exploratory study).

ELIGIBILITY:
Inclusion Criteria:

ALL:

* Informed consent
* Affiliation to social security
* Preliminary medical examination

PATIENTS WITH EPILEPSY:

* Symptomatic drug-resistant anterior temporal epilepsy (confirmed with video-electroencephalography and magnetic resonance imaging and if necessary intracerebral SEEG exploration)
* Patient needing anterior temporal lobectomy and undergoing pre-surgery conventional intercritical assessment for surgery decision
* Nonverbal IQ ≥ 70 (WAIS-IV)
* At least 6 successful VOSP tests (perception test)

Exclusion Criteria:

ALL:

* persons under legal protection or incapable to consent
* Persons deprived of liberty by juridical or administrative decision

PATIENTS WITH EPILEPSY:

- Sever visual disorders of neurological or ophthalmological origin

CONTROL INDIVIDUALS:

* Psychiatric or neurological disorders
* Important ophthalmological disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Scores obtained with Benton test by patients with anterior temporal epilepsy and matched control individuals | day 0

SECONDARY OUTCOMES:
Change of scores obtained with Benton test by epilepsy patients before and after lobectomy and control individuals (only patients having undergone anterior temporal lobectomy and matched control individuals) | day 0 and after 12 to 18 months
Change of scores obtained with Benton test by epilepsy patients before and after lobectomy and control individuals (only patients having undergone anterior temporal lobectomy and matched control individuals) | day 0 and after 24 to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Louis Maillard, Principal Investigator — Service de Neurologie, Hôpital Central, CHU de Nancy, France
Locations (1):
- Service de Neurologie, Hôpital Central, CHU de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No